CLINICAL TRIAL: NCT00493909
Title: Prospective, Randomised, Single-Blinded, Monocentric Clinical Study to Compare Postoperative Analgesia and Outcome After Combined Paravertebral and Intrathecal Versus Thoracic Epidural Analgesia for Thoracotomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital Freiburg (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TL-2007-06
Record Dates: First submitted 2007-06-28; First posted 2007-06-29 (Estimated); Last update posted 2009-02-16 (Estimated); Status verified 2009-02

CONDITIONS: Pain, Postoperative
Keywords: thoracotomy; pain therapy; thoracic paravertebral blockade; intrathecal opioids; thoracic epidural analgesia; Analgesia after thoracotomy
MeSH Terms: conditions — Pain, Postoperative; Agnosia | interventions — Tea

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): thoracic epidural analgesia
  Interventions: Procedure: intrathecal opioids and thoracic paravertebral analgesia; Procedure: thoracic epidural analgesia
- 2 (Active Comparator): intrathecal opioids and thoracic paravertebral analgesia
  Interventions: Procedure: intrathecal opioids and thoracic paravertebral analgesia

INTERVENTIONS:
Procedure: intrathecal opioids and thoracic paravertebral analgesia
Procedure: thoracic epidural analgesia
  Arms: 1

SUMMARY:
The purpose of this study is to compare whether epidural analgesia would provide equal analgesia than combining intrathecal opioids with thoracic paravertebral local anesthetics.

DETAILED DESCRIPTION:
Thoracotomy is an invasive surgical procedure, which is mainly performed in patients with pre-existing lung disease such as lung cancer or chronic obstructive pulmonary disease. Pain after thoracotomy is considered the most intense acute postoperative pain, adversely affecting the ability to cough, deep breathing, and lung function, resulting in respiratory complications and delayed recovery. The adverse effects can be further aggravated by occurrence of chronic post-thoracotomy pain.

Thoracic epidural analgesia is often recommended as the gold standard for the relief of acute post-thoracotomy pain. Thoracic paravertebral blockade or intrathecal opioid analgesia has also been shown to be efficacious for pain relief. Since there is no ideal single regional technique for pain relief after thoracotomy an alternative method maybe the combination of low-dose intrathecal morphine and sufentanil plus continuous thoracic paravertebral analgesia with local anesthetics.

We therefore hypothesized that combining intrathecal sufentanil and morphine with thoracic paravertebral applicated ropivacaine would provide equal analgesia compared to thoracic epidural analgesia with ropivacaine and sufentanil. We further speculate that this new regimen would have a lower incidence of typical side effects due to TEA, such as block failure, hypotension or urinary retention.

ELIGIBILITY:
Inclusion Criteria:

* Sex: male/female
* Age: 18 - 75 years
* Informed consent of the patient
* Elective thoracotomy
* Two chest drains

Exclusion Criteria:

* Contraindications against the use of regional techniques: known allergy to local anesthetics
* Infection around the puncture site
* Coagulation disorders
* Drug abuse
* Emergency surgery
* Pregnancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2007-06; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
The primary outcome measures used are pain at rest, at coughing, and on movement at each time point, as reported by the patient using a standard Visual Analogue Score (VAS). | within the first three days

SECONDARY OUTCOMES:
incidence of side-effects (nausea, vomiting, sedation score, respiratory depression, hypotension, pruritus, urinary retention), total number of doses of piritramide administered, patient satisfaction, and incidence of chronic pain. | within one year

CONTACTS AND LOCATIONS:
Overall Officials: Torsten Loop, M.D., Principal Investigator — Department of Anesthesiology and Critical Care Medicine, University Medical Center, Hugstetterstrasse 55, D-79106 Freiburg, Germany,; Sebastian Dango, M.D., Principal Investigator — Department of Thoracic Surgery, University Medical Center, Hugstetterstrasse 55, D-79106 Freiburg, Germany,
Locations (1):
- Department of Thoracic Surgery, University Medical Center, Freiburg im Breisgau, Germany

REFERENCES:
- [Derived] Dango S, Harris S, Offner K, Hennings E, Priebe HJ, Buerkle H, Passlick B, Loop T. Combined paravertebral and intrathecal vs thoracic epidural analgesia for post-thoracotomy pain relief. Br J Anaesth. 2013 Mar;110(3):443-9. doi: 10.1093/bja/aes394. Epub 2012 Nov 14. PMID 23151421